CLINICAL TRIAL: NCT05173844
Title: E-buddy Supported Digital Sleep Therapy for Older Adults With Cognitive Impairment
Brief Title: Digital Sleep Therapy for Older Adults With Cognitive Impairment
Acronym: ExCEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X21-0434
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-06

CONDITIONS: Insomnia Type; Sleep Disorder; Cognitive Impairment
MeSH Terms: conditions — Sleep Wake Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants will be instructed to use SleepFix mobile application for 3 weeks with an optional 3 weeks of additional therapy. Participants will complete daily sleep diary entries (which take less than 1 min) which are used to calculate the sleep window titration. SleepFix incorporates sleep restriction and stimulus control which have been shown to be the most powerful components of cognitive-behavioural therapy for insomnia - CBTi. It has been shown to produce rapid, clinically-meaningful insomnia symptom reduction in a shorter period of time compared with both face-to-face and digital CBTi. SleepFix does not require the user to complete modules and multiple components such as other digital CBTi programs (e.g. Sleepio). Further, it is personalised to the individual's current sleep patterns and requires minimal engagement compared to full CBTi.
  Interventions: Other: SleepFix mobile application
- Control (No Intervention): Participants randomised to the control group will gain access to the first Sleep Health Education module immediately following completion of baseline questionnaires. There are 3 modules provided bi-weekly and the information in these modules is presented as a subdomain through the study website. The participant will receive a link to this information as each module is made available. Control participants will have full access to these modules for the duration of the study.

INTERVENTIONS:
Other: SleepFix mobile application — Digital behavioural therapy (dBTi) mobile application SleepFix® is specifically designed to treat insomnia and has been shown to be engaging and clinically efficacious.
  Arms: Treatment

SUMMARY:
This study aims to determine the efficacy of digital Behavioural Therapy for Insomnia (dBTi) compared to online sleep health education (control) at reducing insomnia symptom severity (Insomnia Severity Index: ISI) in older adults (50+ years) with subjective cognitive impairment from baseline compared to week 8.

DETAILED DESCRIPTION:
Insomnia is a highly prevalent sleep disorder affecting up to 10% of the adult population and reports of over 40% in the older population. Current insomnia treatments focus heavily on symptom management with cognitive behavioural therapy for insomnia (CBTi), in both digital and face-to-face form as the recommended first-line treatment. Despite the strong evidence for digital CBTi, there are a lack of data related to older people and whether digital brief behavioural therapy is efficacious in this population. Recent work shows that sleep plays a critical role in optimising brain function and sleep disturbance is highly prevalent in individuals with cognitive impairment.

The investigators will conduct a fully online study comparing 3-weeks of digital brief behavioural therapy for insomnia (dBBTi) (in addtiotion to an extra optional 3 weeks) against online sleep health education. Participants will be recruited, screened and determined eligibility and consent will be conducted online. Participants will be randomly allocated to either dBBTi delivered via a mobile application called SleepFix or wait-listed control. The SleepFix mobile application delivers sleep restriction therapy using a 4 stage approach to improve sleep efficiency. The control will consist of 3 online sleep health education modules provided bi-weekly with information about sleep and sleep hygiene without any specific insomnia therapy. Participants will be recruited using social media and directed to a website to determine eligibility and then provided access to either the dBBTi (SleepFix) or the control with a link to the first online module.

At baseline, all participants will complete self-reported measures of insomnia, cognition ,sleep, fatigue, sleepiness , anxiety, depression, quality of life and digital health literacy. These will be repeated at follow-up at weeks 8, 16.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years and older
* Insomnia Severity Index score ≥10
* Self-reported subjective cognitive impairment as defined as moderate subjective cognitive complaints (i.e. answers YES to have cognitive concerns OR thinking and memory skills are worse than same-age peers on the online screening)
* English speaking
* Access to a smartphone and willingness/proficiency to use a mobile app for healthcare
* Able to give informed online consent

Exclusion Criteria:

* Neurological (e.g. Parkinson's, epilepsy) and major psychiatric disease (e.g. current major depression), dementia, history of cerebrovascular events (stroke, TIA); history of head injury with loss of consciousness > 30mins;
* Self-reported jetlag symptoms due to travel in the last 7 days;
* Current illicit substance use or alcohol intake suggestive of a hazardous or harmful pattern;
* Shift-work;
* Medical conditions with known effects on cognition and sleep (e.g. cancer with chemotherapy);
* Diagnosed obstructive sleep apnoea, or other sleep disorder including REM Sleep Behaviour Disorder, Restless Legs Syndrome or Narcolepsy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | Change score from baseline at 8 weeks
  Insomnia Severity Index (ISI) is a 7-item questionnaire used to examine overall insomnia severity. It consists of a five-point Likert type scale for each item (ranging from "no problem" = 0 to "severe problem" = 4) regarding symptoms over the past 2 weeks. Scores range from 0-28 with higher scores indicating greater insomnia symptom severity.

SECONDARY OUTCOMES:
Change in self-reported cognitive impairment | Change score from baseline at 8 weeks
  The British Columbia Cognitive Complaints Inventory (BC-CCI)12 is a 6-item tool to assess self-perceived cognitive decline. It probes any perceived problems associated with cognition, memory, expressive language, word finding, processing speed, and problem solving in reflection of the last 7 days. Answers for each question range from 0 (= "not at all") to 3 (= "Very much"). Scores are summed to a total out of 18 that reflects the cognitive complaint severity. The BC-CCI has a short reference period to ensure that it only reflects complaints outside of the treatment window.
Change in sleep metrics and quality | Change score from baseline at 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-reported questionnaire which assesses sleep quality and disturbances over the previous 2 weeks so only variables across a time-period not including the therapy window are measured. Seven component scores are derived from the responses, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0-21) where a score of 5 or more indicates poor sleep quality.
Change in depressive symptoms | Change score from baseline at 8 weeks
  The Geriatric Depression Scale (GDS) is a self-report measure of depression in older adults. Users respond in a "Yes/No" format. The shortened form comprises of 15 items chosen from the Geriatric Depression Scale-Long Form. These 15 items were chosen because of their high correlation with depressive symptoms in previous validation studies. Of the 15 items, 10 indicate the presence of depression when answered positively while the other 5 are indicative of depression when answered negatively. This form can be completed in approximately 5 to 7 minutes, making it ideal for people who are easily fatigued or are limited in their ability to concentrate for longer periods of time.
Change in anxiety symptoms | Change score from baseline at 8 weeks
  The General Anxiety Disorder-7 (GAD-7) is a 7-item self-administered scale used to assess the severity of generalised anxiety by asking how often participants have experienced symptoms in the previous two weeks. It consists of a three-point Likert type scale for each item (ranging from "not at all" = 0 to "nearly every day" = 3). All items are summed with total scores ranging from 0-21 where 5, 10 and 15 indicate the cut-off scores for mild, moderate and severe anxiety, respectively.
Change in fatigue | Change score from baseline at 8 weeks
  The Flinders Fatigue Scale (FFS) is a 7-item self-reported instrument designed to measure the level of subjective daytime fatigue experienced over the previous two weeks. 6-items consist of a 5-point Likert type scale ranging from "not at all" = 0 to "extremely" = 4. Item 5 uses a multiple-item checklist and is scored as a sum. All items are summed with total scores ranging from 0-31 with higher scores reflecting greater fatigue.
Change in daytime sleepiness | Change score from baseline at 8 weeks
  The Epworth Sleepiness Scale (ESS) is an 8-item self-reported questionnaire that provides a rating of general sleepiness in the last two weeks. Participants are asked to rate each item on a 4-point Likert scale from "would never dose" = 0 to "high chance of dozing" = 3. All items are summed with total scores ranging from 0-26 where scores >10 and >15 reflect above-average and pathological daytime sleepiness, respectively.
Change in quality of Life | Change score from baseline at 8 weeks
  The EuroQol five-dimensional (EQ-5D) is a well-validated, generic instrument for measuring health related quality of life at the time of completion. The self-reported questionnaire is comprised of 2 components including: (1) Health state description - measured in terms of 5 dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression and (2) evaluation - where participants are asked to evaluate their overall health using a visual analogue scale. In Part 1, each item is assigned a level (ranging from "indicating no problem"1 - "indicating unable to/extreme problems" - 5) according to the response and this descriptive data is used to generate a health-related quality of life profile for the subject. Part II is scored from 0 (worst health state imaginable) to 100 (best health state imaginable).
Digital literacy | The questionnaire will only be collected at baseline
  The eHEALS Literacy Scale (eHEALS) will be used to assess digital health literacy. eHEALS is an 8-item, 5-point Likert-type questionnaire that measures a participant's perception of, and ability toward electronic health information27. Responses range from "strongly disagree" =1, to "strongly agree" = 5. Total scores are summed to range from 8 to 40 where lower scores indicate lower self-reported digital health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gordon, PhD, Principal Investigator — Macquarie University
Locations (1):
- Woolcock Institute of Medical Research, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data may be made available upon the Principal investigator's agreement with an amendment required to the approving ethics board.
Supporting Information: Study Protocol, ICF
Time Frame: The study data will be available following all analyses.
Access Criteria: Contact the Coordinating Principal Investigator for access to data.